CLINICAL TRIAL: NCT02602288
Title: Multilevel Tobacco Intervention in Community Clinics for Underserved Families
Brief Title: Babies Living Safe and Smokefree
Acronym: BLiSS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Temple University (Other)
Collaborators: N.O.R.T.H., Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R01CA188813 (NIH)
Record Dates: First submitted 2015-11-09; First posted 2015-11-11 (Estimated); Results first posted 2022-03-15 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-02

CONDITIONS: Second Hand Tobacco Smoke; Nicotine Dependence
MeSH Terms: conditions — Tobacco Use Disorder | interventions — corticosteroid hormone-induced factor; Referral and Consultation; Tobacco Use Cessation Devices; Nicotine Chewing Gum

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AAR+Behavioral Intervention (EXP) (Experimental): Ask Advise Refer (AAR): WIC clinic staff ask about children's secondhand smoke exposure (SHSe), advise about harms of SHSe, and refer to smoking cessation resources. Telebased tobacco counseling: Telephone counseling to promote parent's smoking cessation and behaviors to protect children from secondhand tobacco smoke. Mobile phone smoking cessation application: Smartphone based application to support smoking cessation efforts. Nicotine polacrilex: Over the counter nicotine replacement therapy in gum or lozenge form.
  Interventions: Behavioral: Ask, Advise, Refer; Behavioral: Telebased tobacco counseling; Device: Mobile phone smoking cessation application; Drug: Nicotine polacrilex
- AAR+Attention Control Intervention (CTL) (Active Comparator): Ask Advise Refer (AAR): WIC clinic staff ask about children's secondhand smoke exposure (SHSe), advise about harms of SHSe, and refer to smoking cessation resources. Telebased nutrition counseling: Telephone counseling to promote nutritious eating practices in the family. Mobile phone nutrition application: Smartphone based application to support healthy eating habits
  Interventions: Behavioral: Ask, Advise, Refer; Behavioral: Telebased nutrition counseling; Device: Mobile phone nutrition application

INTERVENTIONS:
Behavioral: Ask, Advise, Refer — WIC clinic staff ask about children's secondhand smoke exposure (SHSe), advise about harms of SHSe, and refer to smoking cessation resources
Behavioral: Telebased tobacco counseling — Telephone counseling to promote parent's smoking cessation and behaviors to protect children from secondhand tobacco smoke
  Arms: AAR+Behavioral Intervention (EXP)
Behavioral: Telebased nutrition counseling — Telephone counseling to promote nutritious eating practices in the family.
  Arms: AAR+Attention Control Intervention (CTL)
Device: Mobile phone smoking cessation application — Smartphone based application to support smoking cessation efforts
  Arms: AAR+Behavioral Intervention (EXP)
Device: Mobile phone nutrition application — Smartphone based application to support healthy eating habits
  Arms: AAR+Attention Control Intervention (CTL)
Drug: Nicotine polacrilex — Over the counter nicotine replacement therapy in gum or lozenge form.
  Other Names: nicotine gum, nicotine lozenge
  Arms: AAR+Behavioral Intervention (EXP)

SUMMARY:
The purpose of this randomized controlled trial is to develop and test the efficacy of a multilevel, multimodal intervention designed to modify maternal smoking behavior to reduce children's exposure to secondhand tobacco smoke (primary outcome) and promote their smoking cessation (secondary outcome). Low-income mothers who smoke will be enrolled. Mothers will be recruited from the supplemental nutrition program, Women, Infants and Children (WIC) clinics. All mothers visiting WIC clinics will receive a clinic-level intervention, which consists of nutrition counselors following an "ask, advise, and refer" protocol to identify if their children are exposed to secondhand tobacco smoke, advise mothers who smoke about the harms of such exposure and the benefits of reducing exposure, and referring mothers to the trial. Screened eligible mothers will be consented and randomized to an attention control condition focused on nutrition (CTL) or to an experimental (EXP) multimodal behavioral intervention that integrates telebased counseling to promote the reduction of child secondhand smoke exposure (SHSE) and maternal smoking with an adjunct smoking cessation mobile app and nicotine replacement therapy use. The investigators will test the primary hypothesis that relative to children in the CTL condition, those in the EXP condition will have lower exposure SHSE as measured by mothers' reports and child cotinine levels. The investigators will also test the secondary hypothesis that relative to mothers in the CTL condition, those in the EXP condition will have higher bioverified 7-day point prevalence quit rates. In addition, the study will: (a) evaluate if specific psychosocial and behavioral factors-- social support, urge coping skills, self-efficacy, and SHSe protective behaviors--mediate the effects of the EXP intervention on outcomes and (b) explore whether other residential smokers, level of nicotine dependence, depressive/anxious symptoms, weight concerns, intervention dosage, and pregnancy status predict outcomes and moderate treatment effects.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* female
* at least 18 years of age
* parent or legal guardian of child under 6 yrs old who lives with them at least 4 days/wk
* smokes

Exclusion Criteria:

* non-nicotine drug dependence
* active psychiatric disturbance (bipolar, schizophrenia, psychosis)
* inadequate health literacy
* pregnant
* no smartphone

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 396 (Actual)
Dates: Start 2016-02; Primary Completion 2019-10-23 (Actual); Study Completion 2019-10-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen J Lepore, PhD, Principal Investigator — Temple University
Locations (2):
- United States (2):
  - Temple University, Philadelphia, Pennsylvania
  - N.O.R.T.H., Inc., Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Collins BN, Lepore SJ, Egleston BL. Eliminating children's tobacco smoke exposure: a pathway to bioverified abstinence among low-income maternal smokers in the Babies Living Safe and Smokefree (BLiSS) trial. J Behav Med. 2023 Dec;46(6):1042-1048. doi: 10.1007/s10865-023-00423-9. Epub 2023 Jun 7. PMID 37285107
- [Derived] Collins BN, Lepore SJ, Egleston BL. Multilevel Intervention for Low-Income Maternal Smokers in the Special Supplemental Nutrition Program for Women, Infants, and Children (WIC). Am J Public Health. 2022 Mar;112(3):472-481. doi: 10.2105/AJPH.2021.306601. PMID 35196033
- [Derived] Lepore SJ, Collins BN, Killam HW, Barry B. Supportive Accountability and Mobile App Use in a Tobacco Control Intervention Targeting Low-Income Minority Mothers Who Smoke: Observational Study. JMIR Mhealth Uhealth. 2021 Jul 2;9(7):e28175. doi: 10.2196/28175. PMID 34255698
- [Derived] Collins BN, Lepore SJ. Babies Living Safe & Smokefree: randomized controlled trial of a multilevel multimodal behavioral intervention to reduce low-income children's tobacco smoke exposure. BMC Public Health. 2017 Mar 14;17(1):249. doi: 10.1186/s12889-017-4145-7. PMID 28288601

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Nutrition professionals at 10 of Philadelphia's Women, Infants and Children (WIC) clinics conducted the Ask, Advise, Refer protocol to refer women to the study from February of 2016 to October of 2018.
Pre-assignment Details: A total of 2846 women were referred to the trial: 788 were not eligible, 647 were never reached for screening, and 709 declined to be screened. Of 702 that screened eligible, 104 refused consent and 202 could not be reached for consent or baseline. A total of 396 participants were randomized between the two arms of the study.
Period: End of Treatment/3 Month Follow-up
Arm/Group | AAR+Behavioral Intervention (EXP) | AAR+Attention Control Intervention (CTL)
Started | 199 | 197
Completed | 174 | 179
Not Completed | 25 | 18
Not completed — Lost to Follow-up | 14 | 10
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Withdrawn - refused treatment | 9 | 6
Period: 12 Month Follow-up
Arm/Group | AAR+Behavioral Intervention (EXP) | AAR+Attention Control Intervention (CTL)
Started | 174 | 179
Completed | 172 | 175
Not Completed | 2 | 4
Not completed — Lost to Follow-up | 0 | 4
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AAR+Behavioral Intervention (EXP) | AAR+Attention Control Intervention (CTL) | Total
Number analyzed (Participants) | 199 | 197 | 396
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.81 (6.40) | 30.42 (6.64) | 30.11 (6.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 199 | 197 | 396
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 31 | 29 | 60
  Not Hispanic or Latino | 168 | 168 | 336
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 142 | 138 | 280
  White | 26 | 30 | 56
  More than one race | 13 | 11 | 24
  Unknown or Not Reported | 18 | 18 | 36
Region of Enrollment [Number; unit: participants]
  United States | 199 | 197 | 396
Living with spouse/partner [Count of Participants; unit: Participants] | 74 | 72 | 146
High school diploma or less [Count of Participants; unit: Participants] | 124 | 119 | 243
Other smokers live in home [Count of Participants; unit: Participants] | 100 | 98 | 198
Have smoking restrictions in home [Count of Participants; unit: Participants] | 171 | 176 | 347
Average cigarettes smoked per day [Mean (Standard Deviation); unit: cigarettes smoked per day] | 8.83 (5.63) | 8.94 (5.24) | 8.89 (5.43)
Child (log) cotinine [Mean (Standard Deviation); unit: log transformed ng/mL] | .98 (.65) | .97 (.59) | .97 (.62)
Problem drinker on TWEAK scale [Count of Participants; unit: Participants] — The TWEAK alcohol screening test is a short, five-question test that was originally designed to screen pregnant women for harmful drinking habits. The name of the test is an acronym for tolerance, worried, eye-opener, amnesia, and k/cut down (with a poetic license use of "K" instead of "C" for cutting down on alcohol consumption). A total score of two or more on the test is an indication of harmful drinking and further evaluation is indicated.
  Participants | 25 | 12 | 37
Meets depression cutoff on CESD [Count of Participants; unit: Participants] — A score greater than or equal to 10 indicates significant distress or a positive screen for depression.
  Participants | 90 | 89 | 179

OUTCOME MEASURES:

1. Primary Outcome: Child Urine Cotinine
Description: Child urine cotinine is a biomarker for assessing secondhand smoke exposure. The investigators anticipate the EXP group will evidence a greater reduction in child urine cotinine over time than the CTL group. Cotinine values were log transformed to normalize distributions.
Time Frame: 3 months and 12 months
Population: At 12 month follow-up the greater number of units analyzed compared to participants analyzed in the treatment group relates to increased participant compliance with providing a urine sample. At all timepoints the fewer number of cotinines collected compared to self-report data reflects non-compliance among some participants to provide a urine sample following the telephone self-report assessments.
Measure: Mean (Standard Deviation); unit: log transformed ng/mL
Arm/Group | AAR+Behavioral Intervention (EXP) | AAR+Attention Control Intervention (CTL)
Number analyzed (Participants) | 168 | 174
log transformed ng/mL
  3 month follow-up: number analyzed (Participants) | 166 | 174
  3 month follow-up | 1.00 (0.67) | .97 (.63)
  12 month follow-up: number analyzed (Participants) | 168 | 172
  12 month follow-up | 1.09 (0.73) | 1.00 (0.68)

2. Primary Outcome: Cigarettes/Day
Description: Parental report of cigarettes child is exposed to each day in the home and car and other locations by all sources during the 7 days prior to assessment. The investigators anticipate the EXP group will evidence greater reductions in child secondhand smoke exposure over time than the CTL group.
Time Frame: 3 months and 12 months
Population: The lower number of participants analyzed for this item compared to the number of participants completing this assessment battery is due to non-compliance in completing this item among some participants.
Measure: Mean (Standard Deviation); unit: Cigarettes/day secondhand smoke exposure
Arm/Group | AAR+Behavioral Intervention (EXP) | AAR+Attention Control Intervention (CTL)
Number analyzed (Participants) | 172 | 178
Cigarettes/day secondhand smoke exposure
  3 month follow-up | 3.00 (4.89) | 4.47 (6.08)
  12 month follow-up: number analyzed (Participants) | 170 | 173
  12 month follow-up | 3.03 (5.14) | 3.81 (5.04)

3. Secondary Outcome: Parent-reported Cotinine-verified 7-day Point Prevalence Abstinence
Description: When a participant reports smoking abstinence, the investigators will bioverify their smoking status.
Time Frame: 7 days prior to 3 month and 12 month assessments
Population: The number of participants analyzed reflects number of people completing assessment plus recoding participants who were lost to follow up as 0 = not quit.
Measure: Count of Participants; unit: Participants
Arm/Group | AAR+Behavioral Intervention (EXP) | AAR+Attention Control Intervention (CTL)
Number analyzed (Participants) | 174 | 179
Participants
  3 month follow-up | 14 | 2
  12 month follow-up: number analyzed (Participants) | 172 | 175
  12 month follow-up | 15 | 7

ADVERSE EVENTS:
Time Frame: Adverse events were tracked for each participant (enrolled mothers) from the time of the baseline assessment through the 12-month assessment.
Groups:
- AAR+Behavioral Intervention (EXP): Ask. Advise. Refer (AAR): WIC clinic staff ask mothers about children's secondhand smoke exposure (SHSe), advise about harms of SHSe, and refer to smoking cessation resources. Telebased tobacco counseling: Telephone counseling to promote parents' smoking cessation and behaviors to protect children from secondhand tobacco smoke. Mobile phone smoking cessation application: Smartphone-based application to support smoking cessation efforts. Nicotine polacrilex: Over-the-counter nicotine replacement therapy in gum or lozenge form.
  Ask, Advise, Refer: WIC clinic staff ask about children's secondhand smoke exposure (SHSe), advise about harms of SHSe, and refer to smoking cessation resources
  Telebased tobacco counseling: Telephone counseling to promote parent's smoking cessation and behaviors to protect children from secondhand tobacco smoke
  Mobile phone smoking cessation application: Smartphone based application to support smoking cessation efforts
  Nicotine polacrilex: Over the counter nicotine replacement therapy in gum or lozenge form.
- AAR+Attention Control Intervention (CTL): Ask. Advise. Refer (AAR): WIC clinic staff ask mothers about children's secondhand smoke exposure (SHSe), advise about harms of SHSe, and refer to smoking cessation resources. Telebased nutrition counseling: Telephone counseling to promote nutritious eating practices in the family. Mobile phone nutrition application: Smartphone-based application to support healthy eating habits
  Ask, Advise, Refer: WIC clinic staff ask about children's secondhand smoke exposure (SHSe), advise about harms of SHSe, and refer to smoking cessation resources
  Telebased nutrition counseling: Telephone counseling to promote nutritious eating practices in the family.
  Mobile phone nutrition application: Smartphone based application to support healthy eating habits
Arm/Group | AAR+Behavioral Intervention (EXP) | AAR+Attention Control Intervention (CTL)
All-Cause Mortality (participants affected / at risk) | 0/199 | 0/197
Serious Adverse Events (participants affected / at risk) | 0/199 | 0/197
Other Adverse Events (participants affected / at risk) | 0/199 | 0/197

LIMITATIONS AND CAVEATS:
Limited generalizability of findings due to high rates of ineligibility (27.7%) and inability to contact (22.7%) among maternal smokers referred to the trial by WIC nutrition professionals who provided the clinic-level intervention.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2015-12-15): https://cdn.clinicaltrials.gov/large-docs/88/NCT02602288/Prot_SAP_ICF_000.pdf